CLINICAL TRIAL: NCT05152589
Title: Newborn Hearing Loss
Brief Title: Maternal Diabetes in Newborns With Hearing Loss
Acronym: GDM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-21-1070
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Gestational Diabetes; Pregestational Diabetes; Hearing Loss
MeSH Terms: conditions — Diabetes, Gestational; Hearing Loss | interventions — Hearing Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- gestational diabetic mother: Hearing tests of the babies of pregnant women who are being followed up with the diagnosis of gestational diabetes in the peritanotogy clinic
  Interventions: Diagnostic Test: hearing test
- pregestational diabetic mother: Hearing tests of the babies of pregnant women who are being followed up with the diagnosis of pregestational diabetes in the peritanotogy clinic
  Interventions: Diagnostic Test: hearing test
- non diabetic mother: Hearing tests of babies whose mothers do not have gestational or pregestational diabetes
  Interventions: Diagnostic Test: hearing test

INTERVENTIONS:
Diagnostic Test: hearing test — Auditory Brainstem Response (ABR) Test
  Other Names: ABR

SUMMARY:
This study aims to investigate the presence and characteristics of maternal diabetes as a risk factor in newborns with hearing loss.

Hearing loss is one of the most common congenital anomalies among newborns. The newborn hearing screening program is important for early diagnosis in newborns with hearing loss.Gestational diabetes, on the other hand, is a metabolic disease that occurs during pregnancy and can cause complications as in other diabetes mellitus patients.

Despite our knowledge of major complications, the effect of the hyperglycemic intrauterine environment on hearing outcomes has not been adequately studied. The inner ear does not store energy, so it has a particularly high sensitivity to altered blood sugar and insulin. Altered inner ear metabolism leads to auditory and balance disorders.

There is no study in the literature comparing uncomplicated gestational diabetes and pregestational diabetes as a prenatal complication that poses a risk of hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* POSTNATAL AGE BETWEEN 0-28 DAYS
* BIRTH WEIGHT ≥2000GR
* TO HAVE TESTED ON THE NEWBORN HEARING SCREENING UNIT AT ANKARA CITY HOSPITAL

Exclusion Criteria:

* PRETERMS
* CRANIOFACIAL ANOMALIES
* INTRAUTERINE INFECTIONS
* BIRTH WEIGHT <2000 GR

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: NEWBORNS WHO CANNOT PASS THE HEARING TEST APPLIED AS ROUTINE SCREENING
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Hearing Loss | 6 months
  Hearing test results in babies with no diabetes, pregestational diabetes, and gestational diabetes

SECONDARY OUTCOMES:
diabetic mother | 6 months
  Evaluation of classification tests by separating them from subgroups according to mothers' control times, usage controls, and glycemic viewers

CONTACTS AND LOCATIONS:
Locations (1):
- Fuat Emre Canpolat, Ankara, [Select], Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No